CLINICAL TRIAL: NCT02394093
Title: An Open Label Crossover Pharmacokinetic Trial of Aspirin Dry Powder Versus Aspirin Tablets and Aspirin Effervescent Tablets in Healthy Adult Subjects
Brief Title: To Evaluate the Bioavailability of a Single Oral Dose of the Acetylsalicylic Acid Containing Dry Powder 500 mg in Comparison to the Bioavailability of a Single Oral Dose of Aspirin Tablets and Aspirin Effervescent Tablets in Healthy Adults.
Acronym: Icicle
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 17494
Record Dates: First submitted 2015-03-14; First posted 2015-03-20 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-09

CONDITIONS: Pharmacology, Clinical
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aspirin dry powder (Experimental): 500 mg Acetylsalicylic Acid (ASA) dry powder
  Interventions: Drug: Aspirin (Acetylsalicylic acid, BAYe4465)
- Aspirin coated tablet (Active Comparator): 500 mg ASA coated tablet
  Interventions: Drug: Aspirin (Acetylsalicylic acid, BAYe4465)
- Aspirin effervescent tablet (Active Comparator): 500 mg ASA effervescent tablet
  Interventions: Drug: Aspirin (Acetylsalicylic acid, BAYe4465)

INTERVENTIONS:
Drug: Aspirin (Acetylsalicylic acid, BAYe4465) — One stick pack containing 500 mg acetylsalicylic acid dry powder
  Arms: Aspirin dry powder
Drug: Aspirin (Acetylsalicylic acid, BAYe4465) — One tablet containing 500 mg acetylsalicylic acid
  Arms: Aspirin coated tablet
Drug: Aspirin (Acetylsalicylic acid, BAYe4465) — One effervescent tablet containing 500 mg acetylsalicylic acid
  Arms: Aspirin effervescent tablet

SUMMARY:
To evaluate the bioavailability of a single oral dose of the Acetylsalicylic Acid containing dry powder 500 mg in comparison to the bioavailability of a single oral dose of aspirin tablets and aspirin effervescent tablets in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy ,male and female subjects 18 to 55 years of age, inclusive
* Body Mass Index (BMI) of approximately 18 to 30 kg/m2, and a total body weight >50 kg (110 lbs)
* Results of screening and clinical laboratory tests are within normal limits or considered not clinically significant by the Principal Investigator or Sponsor
* Female subjects of childbearing potential must be using a medically acceptable form of birth control for at least 1 month prior to screening (3 months on oral contraceptives), e.g., oral or patch contraceptives, intrauterine device, intramuscular injection or double-barrier and have a negative pregnancy test at Screening and on Day 0 of each treatment period. Female subjects of nonchildbearing potential must be amenorrheic for at least 2 years or had a hysterectomy and/or bilateral oophorectomy.

Exclusion Criteria:

* History of hypersensitivity to acetylsalicylic acid (ASA), naproxen sodium, acetaminophen, other non-steroidal anti-inflammatory drugs (NSAIDs), and similar pharmacological agents or components of the products
* History of gastrointestinal bleeding or perforation, including bleeding related to previous NSAID therapy. Active, or history of recurrent peptic ulcer/hemorrhage (two or more distinct episodes of proven ulceration or bleeding).
* Have taken ASA, ASA-containing products, acetaminophen or any other NSAID (OTC or prescription) seven days prior to dosing or during the Treatment Periods, other than study product
* Loss of blood in excess of 500 mL within 56 days of the first dose of trial treatment (e.g., donation, plasmapheresis, or injury)
* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic disease, or malignancies
* Positive alcohol or drug screen at Screening or on Day 0 of Treatment Periods 1,2 and 3
* Females who are pregnant or lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2015-02; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of Acetylsalicylic Acid (ASA) characterized by AUC0-t | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
Plasma concentration of Acetylsalicylic Acid (ASA) characterized by AUC0-∞ | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
  AUC0-∞ : AUC from zero to infinity after single dose.
Plasma concentration of Acetylsalicylic Acid (ASA) characterized by Cmax | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
  Cmax: maximum drug concentration in plasma after single dose administration
Plasma concentration of Acetylsalicylic Acid (ASA) characterized by tmax | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
  tmax: time to reach maximum drug concentration in plasma after single (first) dose
Plasma concentration of Acetylsalicylic Acid (ASA) characterized by λz (Kel) | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose
  λz (Kel) : Apparent terminal rate constant, calculated from the slope of a log-linear regression of the unweighted data considering the last concentration-time points > LLOQ
Plasma concentration of Acetylsalicylic Acid (ASA) characterized by t1/2 | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
Plasma concentration of Acetylsalicylic Acid (ASA) characterized by t lag | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
  t lag : Lag-time (time delay between drug administration and first observed concentration above LLOQ (Lower limit of quantification)
Plasma concentration of Acetylsalicylic Acid (ASA) characterized by Cmax/AUC0-∞ | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
Plasma concentration of Acetyl salicylic Acid (ASA) characterized by MRT | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
  MRT :Mean residence time (for extravascular and iv bolus administration)
Plasma concentration of Salicylic Acid (SA) characterized by AUC0-t | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
Plasma concentration of Salicylic Acid (SA) characterized by AUC0-∞ | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
  AUC0-∞ : AUC from zero to infinity after single dose
Plasma concentration of Salicylic Acid (SA) characterized by Cmax | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
  Cmax: maximum drug concentration in plasma after single dose administration
Plasma concentration of Salicylic Acid (SA) characterized by tmax | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
  tmax: time to reach maximum drug concentration in plasma after single (first) dose
Plasma concentration of Salicylic Acid (SA) characterized by λz (Kel) | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
  λz (Kel) : Apparent terminal rate constant, calculated from the slope of a log-linear regression of the unweighted data considering the last concentration-time points > LLOQ
Plasma concentration of Salicylic Acid (SA) characterized by t1/2 | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
Plasma concentration of Salicylic Acid (SA) characterized by t lag | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
  t lag : Lag-time (time delay between drug administration and first observed concentration above LLOQ
Plasma concentration of Salicylic Acid (SA) characterized by Cmax/AUC0-∞ | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
Plasma concentration of Salicylic Acid (SA) characterized by MRT | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
  MRT :Mean residence time (for extravascular and iv bolus administration)
Plasma concentration of Acetylsalicylic Acid (ASA) characterized by AUC0-t /AUC0-∞ | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.
Plasma concentration of Salicylic Acid (SA) characterized by AUC0-t /AUC0-∞ | baseline (pre-dose), 5, 7.5, 10, 12.5, 15, 17.5, 20, 22.5, 25, 27.5, 30, 32.5, 35, 37.5, 40, 42.5, 45, 50, 55 minutes and 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 7, 9, 12 and 24 hours post-dose.

SECONDARY OUTCOMES:
Number of participants with Adverse Events as measure of safety and tolerability | Up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Hackensack, New Jersey, United States